CLINICAL TRIAL: NCT02418546
Title: Electronic-health Application To Measure Outcomes REmotely Clinical Trial
Acronym: EAT MORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Anne-Marie Alexandra Wills, MD, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015P000258
Record Dates: First submitted 2015-04-06; First posted 2015-04-16 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Neurodegenerative Disease; Weight Loss; Amyotrophic Lateral Sclerosis; Parkinson's Disease; Huntington's Disease; Cachexia
MeSH Terms: conditions — Neurodegenerative Diseases; Weight Loss; Amyotrophic Lateral Sclerosis; Parkinson Disease; Huntington Disease; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- In-Person Nutritional Counseling (Active Comparator): Participants in the in-person nutritional counseling arm will meet with a Registered Dietitian at every clinic visit and will also receive regular phone calls to monitor weight and food intake. Participants' individual dietary needs will be calculated using baseline calorie consumption, weight history, disease status and current activity level.
  Interventions: Behavioral: In-Person Nutritional Counseling by a Registered Dietitian
- E-Health App for Nutritional Counseling (Experimental): Participants randomized to the e-Health App arm with receive nutritional counseling using the e-Health Application. Participants will enter weights at home and complete electronic food records using the App. Participants' individual dietary needs will be calculated using baseline calorie consumption, weight history, disease status and current activity level. Participants will receive these calorie recommendations through the Application.
  Interventions: Behavioral: Nutritional counseling using an e-Health Application
- Standard Care (No Intervention): Participants are allowed to receive all usual treatments and medications. Participation in other research studies is allowed.

INTERVENTIONS:
Behavioral: In-Person Nutritional Counseling by a Registered Dietitian
  Arms: In-Person Nutritional Counseling
Behavioral: Nutritional counseling using an e-Health Application
  Arms: E-Health App for Nutritional Counseling

SUMMARY:
This is a phase II feasibility, safety, tolerability and preliminary efficacy study of an e-Health application versus in-person nutritional counseling to maintain or increase weight in patients with neurodegenerative diseases including amyotrophic lateral sclerosis (ALS), Parkinson's Disease (PD) and Huntington's disease (HD). Primary Objectives include the feasibility, safety, tolerability and efficacy of an e-Health application to maintain or increase body weight compared to in-person nutritional counseling. Secondary Objectives are to measure the number of calories required to maintain or increase body weight in neurodegenerative diseases at all stages of the disease. Tertiary Objectives are to test the effects of an e-Health application compared to in-person nutritional counseling on disease progression using the ALSFRS-R, UHDRS or UDysRS, on survival, and on quality of life using the PROMIS SF v1.1 scale.

DETAILED DESCRIPTION:
This is a single center, randomized, open-label, placebo controlled, parallel group study. The study treatment period is approximately 6 months and observation period is approximately 7 months. There are three parallel treatment groups: in-person nutritional counseling, nutritional counseling using an e-Health App, and standard care. Subjects will be randomly assigned in a 1:1:1 ratio using a computer-generated randomization scheme. Subjects in the two intervention arms will be given caloric recommendations designed to cause weight stability or modest weight gain, depending on their current BMI and weight loss history. All participants in the intervention arms will receive counseling either in-person or remotely through the App by registered dietitians (RD) working in the Bionutrition department of the Clinical Research Center at MGH. At MGH, approximately 150 ALS subjects (50 per treatment group) will be enrolled. Approximately 75-150 PD and HD subjects will enroll.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with neurodegenerative diseases such as ALS, PD or HD with or without a history of unintentional weight loss.
2. Male or female subjects aged 18 years or older.
3. Participants must be capable of providing informed consent and complying with trial procedures.
4. Participants must have an MGH swallowing screening tool score>5 at the time of the screening visit
5. Participants or a designated caregiver must be able to obtain home weights and communicate to their RD

Exclusion Criteria:

1. Clinical evidence of unstable medical or psychiatric illness, in the investigator's judgment, which would prevent the participant from completing their assessments.
2. BMI > 35 combined with a history of cardiovascular disease; or a history of diabetes regardless of BMI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Wills, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wills AM, Garry J, Hubbard J, Mezoian T, Breen CT, Ortiz-Miller C, Nalipinski P, Sullivan S, Berry JD, Cudkowicz M, Paganoni S, Chan J, Macklin EA. Nutritional counseling with or without mobile health technology: a randomized open-label standard-of-care-controlled trial in ALS. BMC Neurol. 2019 May 29;19(1):104. doi: 10.1186/s12883-019-1330-6. PMID 31142272

RESULTS

PARTICIPANT FLOW:
Groups:
- In-Person Nutritional Counseling: Participants in the in-person nutritional counseling arm will meet with a Registered Dietitian at every clinic visit and will also receive regular phone calls to monitor weight and food intake. Participants' individual dietary needs will be calculated using baseline calorie consumption, weight history, disease status and current activity level.
  In-Person Nutritional Counseling by a Registered Dietitian
- E-Health App for Nutritional Counseling: Participants randomized to the e-Health App arm with receive nutritional counseling using the e-Health Application. Participants will enter weights at home and complete electronic food records using the App. Participants' individual dietary needs will be calculated using baseline calorie consumption, weight history, disease status and current activity level. Participants will receive these calorie recommendations through the Application.
  Nutritional counseling using an e-Health Application
Period: Overall Study
Arm/Group | In-Person Nutritional Counseling | E-Health App for Nutritional Counseling | Standard Care
Started | 26 | 26 | 26
Completed | 19 | 20 | 23
Not Completed | 7 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Person Nutritional Counseling | E-Health App for Nutritional Counseling | Standard Care | Total
Number analyzed (Participants) | 26 | 26 | 26 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.9) | 54.7 (11.5) | 57.5 (10.9) | 56.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 15 | 31
  Male | 16 | 20 | 11 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 25 | 25 | 24 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 26 | 26 | 78
ALS Functional Rating Scale-Revised [Mean (Standard Deviation); unit: Total score in points] — Total score 0-40 with higher scores signifying better function
  Total score in points | 34.9 (6.67) | 37.4 (6.19) | 36.7 (5.36) | 36.4 (6.21)

OUTCOME MEASURES:

1. Primary Outcome: Estimated Mean Change in Weight From Baseline to 6 Months
Description: The Primary Aim is to study the feasibility and efficacy to maintain or increase body weight of an e-Health application and in-person nutritional counseling compared to standard of care and to each other. Weights were measured in the clinic every 3 months.
Time Frame: Change over time from Baseline to 6 months
Population: Please note that these are Parameter Estimates rather than "means"
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | In-Person Nutritional Counseling | E-Health App for Nutritional Counseling | Standard Care
Number analyzed (Participants) | 26 | 26 | 26
kg | -0.1 [-2.1 to 2.0] | -0.2 [-2.4 to 2.1] | -1.2 [-3.2 to 0.7]

2. Secondary Outcome: Change in Calorie Intake Over Time
Description: Secondary aims include measuring the number of calories required to maintain or increase body weight in patients with neurodegenerative diseases. Total daily energy intake was calculated using 4 day food records at baseline, 3 months and 6 months
Time Frame: Change from baseline over 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Safety: Frequency of Adverse Events
Description: To study the safety of an e-Health application and in-person nutritional counseling compared to standard of care and to each other.
Time Frame: From baseline to month 7 (one month after 6 month end of study visit)
Reporting Status: Not Posted

4. Secondary Outcome: Tolerability: The Number of Participants Who Complete the Study While Complying With at Least 80% of the Counseling Sessions
Time Frame: Baseline, 3 months and 6 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Exploratory Efficacy Measure: Survival
Description: Vital status will be measured until the last subject last visit.
Time Frame: baseline to 18 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Exploratory Efficacy Measure: Disease Progression in ALS Functional Rating Scale-Revised (ALSFRS-R)
Description: Disease progression will be measured using disease-specific outcome measures (the ALSFRS-R scale). The range of the ALSFRS-R is 0-40 with higher scores indicating better function. Change in ALSFRS-R is reported as units/month.
Time Frame: Change over time from Baseline to 6 months
Population: Change over time of continuous, longitudinal measures was analyzed using a shared-baseline, mixed effect model with fixed effects for visit and an interaction between post-baseline visit and study arm and with a random slope and intercept for each subject with unstructured covariance.
Measure: Mean (95% Confidence Interval); unit: units per month
Arm/Group | In-Person Nutritional Counseling | E-Health App for Nutritional Counseling | Standard Care
Number analyzed (Participants) | 26 | 26 | 26
units per month | -5.8 [-8.2 to -3.4] | -2.6 [-5.1 to -0.1] | -5.2 [-7.6 to -2.9]

7. Other Pre Specified Outcome: Exploratory Efficacy Measure: Quality of Life
Description: Quality of life will be measured using the PROMIS SF 1.1 in units.
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | In-Person Nutritional Counseling | E-Health App for Nutritional Counseling | Standard Care
All-Cause Mortality (participants affected / at risk) | 4/26 | 0/26 | 1/26
Serious Adverse Events (participants affected / at risk) | 4/26 | 5/26 | 2/26
Other Adverse Events (participants affected / at risk) | 9/26 | 11/26 | 12/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Person Nutritional Counseling (N=26) | E-Health App for Nutritional Counseling (N=26) | Standard Care (N=26)
Deep Venous Thrombosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ewing's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-Person Nutritional Counseling (N=26) | E-Health App for Nutritional Counseling (N=26) | Standard Care (N=26)
sialorrhea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1)
Falls (Injury, poisoning and procedural complications) | 7 (8) | 9 (13) | 9 (13)
Choking (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT02418546/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02418546/SAP_001.pdf